CLINICAL TRIAL: NCT06464783
Title: Effectiveness of Comprehensive Corrective Exercise Program on Kyphosis in Recreational Cyclists
Brief Title: Effectiveness of Comprehensive Corrective Exercises Program on Kyphosis in Recreational Cyclists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: REC/01822 M Khalil Ur Rehman
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Thoracic Kyphosis; Cyclists
Keywords: Comprehensive corrective; Thoracic Flexion; Thoracic Extension; Side flexion; Kyphosis Angle

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive Corrective Exercise Program (Experimental): Comprehensive Corrective Exercise Program includes following exercises.
  Corrective Exercises+ Core strengthening exercises include Chin tuck Supine bridging on stable surface supine bridging with knee flexed on unstable surface unilateral lifting of arms and legs in crawling position Activation of transverse abdominous muscle. Unilateral arms and legs movements in siting position on unstable surface (ball) Cat and camel exercises Contralateral arms and legs movements in siting position on unstable surface (ball)
  Stretching include Stretching of neck extensor muscle Stretching of pectoral muscle group in standing and supine position
  Interventions: Other: Comprehensive Corrective Exercise Program
- Thoracic Exercise Program (Active Comparator): Thoracic Exercise Program includes following exercises.
  Extension exercises include Thoracic extension in kneeling position T W Y I thoracic exercise in prone position.
  Mobilization includes Self-mobilization
  Stretching includes Stretching of pectoral muscle group in standing and supine position
  Interventions: Other: Thoracic Exercise Program

INTERVENTIONS:
Other: Comprehensive Corrective Exercise Program — Week 1st to 2nd: Corrective exercises +Core strengthening (2 sets 10 reps). Stretchings (30 sec hold, 3 reps).
  Week 3rd to 5th: Corrective exercises +Core strengthening (3 sets 15 reps). Stretchings (30 sec hold, 3 reps).
  Week 5th to 8th: Corrective exercises +Core strengthening (3 sets 20 reps). Stretchings (30 sec hold, 3 reps).
  Arms: Comprehensive Corrective Exercise Program
Other: Thoracic Exercise Program — Week 1st to 2nd: Thoracic extension (2 sets 10 reps). Mobilization (60 sec 2 reps). Stretching (30 sec hold and 3 reps).
  Week 3rd to 5th: Thoracic extension (2 sets 15 reps). T W Y I thoracic exercise in prone (2 sets 15 reps). Self-mobilization (60 seconds 2 reps). Stretching (30 sec hold and 3 reps)
  Week 5th to 8th. Thoracic extension (3 sets 20 reps). T W Y I thoracic exercise in prone position (3 sets 20 reps). Self-mobilization (60 sec 2 reps). Stretching (30 sec hold and 3 reps)
  Arms: Thoracic Exercise Program

SUMMARY:
My study aim to investigate the effectiveness of comprehensive corrective exercise program on kyphosis in recreational cyclists. Additionally, i want to investigate the post exercise effects on thoracic kyphosis angle, pain levels and thoracic ranges of motion. Our study on kyphosis in cyclists and what treatment plan could be best to minimize and treat the conditions which are affecting cyclist posture, daily life quality this is very rare study as there are no studies which explains such parameters, in these studies we will effectively describe comprehensive exercise plan to reduce kyphosis angle, increase thoracic roms, decrease pain levels and maintain good quality of life.

DETAILED DESCRIPTION:
Sagittal plane deformity, another name for excessive thoracic spine curvature, is a postural condition marked by an unnatural increase in the thoracic kyphosis angle. This angle typically falls between 20° and 40°, but values of 45° to 50° or higher are thought to be suggestive of hyperkyphosis, increased kyphosis, or postural kyphosis. Because of spinal misalignment, excessive upper back curvature, or hyperkyphosis, can happen at any age.

Athletes are becoming increasingly concerned about kyphosis, an excessive forward curvature of the upper spine, particularly those who play sports like cycling that require a forward-leaning posture. Continuously hunching over the handlebars for extended periods when cycling can exacerbate this condition and result in discomfort, pain, and other problems. Long-term cycling postures can increase the risk of developing kyphosis by causing muscle imbalances, decreased spinal flexibility, and altered biomechanics. In addition to impairing athletic performance, these problems can result in chronic musculoskeletal disorders if left untreated. Sports medicine specialists and physiotherapists need to understand and treat kyphosis in cyclist's top priority as cycling becomes more and more popular. Sports requiring a forward-leaning stance, like swimming, cycling, and some track events, are more likely to cause kyphosis. Because cycling involves postural demands that can result in muscle imbalances and adaptations that increase the risk of kyphosis, cyclists are particularly vulnerable. In this context, the specific postural requirement of cycling includes forward leaning which is crucial for manageability and speed; in relation to kyphosis, this expresses a high degree of causality. This is especially evident during the long training sessions and the continued forward-leaning position in long bike rides that puts a constant stress on the thoracic spine leading to muscle imbalances and hardness in the thoracic region.

Corrective exercise can be defined as exercise that is designed to counter the effects of poor posture and can be effectively done by following the corrective exercise protocol that was created by the National Academy of Sports Medicine (NASM) and has been proven to reduce forward head posture and enhance cervical proprioception which in turn will enhance the general spinal stability. Corrective exercise is needed in fixing postural and musculoskeletal problems. It is a comprehensive process that involves using one's hands to assess muscles and joints, especially for strength and weakness, evaluating one's posture and movement, and prescribing specific exercise regimens to help a client achieve the proper body positioning and function. Corrective exercise training is an advanced method that incorporates ways to avoid overused muscles, stretch short muscles, recruit weak muscles, and embed new movement patterns with the purpose of identifying movement dysfunctions. Besides, it is used in the rehabilitation, conditioning, and performance enhancement training for various impairments that may affect the body regions and flexibility, strength, neuromuscular coordination, and balance. Corrective exercise is an all-inclusive solution for individuals which addresses movement dysfunctions and assist in achieving the maximum physical capability and performance of an individual without causing injury.

ELIGIBILITY:
Inclusion Criteria:● All male recreational cyclist aged below 40

* Cyclists who are riding 1 to 2 hours per day minimum 3 days per week
* Cyclists who have been cycling for at least 2 years.

Exclusion Criteria:

* • All females

  * Elite or master category cyclists
  * Any spinal disorder or recent spinal pain or surgery
  * Any bone pathology or deformity
  * Any musculoskeletal injury
  * Any postural changes due to occupational work setup

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Thoracic Kyphosis Angle | 4th week
  thoracic spine curvature, is a postural condition marked by an unnatural increase in the thoracic kyphosis angle. This angle typically falls between 20° and 40°, but values of 45° to 50° or higher are thought to be suggestive of hyperkyphosis, increased kyphosis, or postural kyphosis.

SECONDARY OUTCOMES:
Visual Analogue Scale | 4th week
  The 10 cm visual analogue scale (VAS), that varies from 0 to 10 and 0 represents "no pain" to 10 as "worst pain imaginable," was used to measure the primary effectiveness outcome based on self-reported pain levels
Thoracic Ranges of motions | 4th week
  Normal values of Thoracic Ranges of motions are as in Thoracic Flexion 50 degrees , thoracic extension 45 degrees, Side Flexion 40 degrees, and thooracic rotation 30 degrees

CONTACTS AND LOCATIONS:
Overall Officials: Waqar ahmed awan, Phd, Study Chair — Riphah International University
Locations (1):
- Kulsum International Hospital Islamabad, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No